CLINICAL TRIAL: NCT02625129
Title: Determining the Clinical Effectiveness and Patient Satisfaction of a Pharmacist-managed Travel Medicine Clinic Under an Expanded Scope of Practice
Brief Title: Effectiveness of and Satisfaction With a Pharmacist-managed Travel Medicine Clinic
Status: Completed | Type: Observational
Sponsor: University of Waterloo (Other)
Collaborators: University of Mississippi Medical Center (Other); Travel Health Network (Other)
Responsible Party: Sponsor
Other Study IDs: 21080
Record Dates: First submitted 2015-11-25; First posted 2015-12-09 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Travel Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pharmacist-provided travel care
  Interventions: Other: Pharmacist-provided travel care

INTERVENTIONS:
Other: Pharmacist-provided travel care — Subjects will receive a pre-travel consultation from a pharmacist with specialty training in travel medicine, and with authorization to prescribe medications and vaccines and administer injections

SUMMARY:
This study will evaluate the clinical effectiveness of, and patient satisfaction with, pre-travel consultations provided by a pharmacist with specialty training in travel medicine and the authorization to prescribe medications and administer vaccinations.

DETAILED DESCRIPTION:
The study will be conducted at the Travel Health Network, a full-service travel medicine clinic located in St. Albert, Alberta. Care will be provided by a pharmacist with a specialized practice in travel medicine, authorization to prescribe vaccines and prescription drugs, and authorization to administer vaccines by injection.

The study will be a prospective mixed-methods cohort study, describing patients receiving care from a pharmacist-managed travel medicine clinic and their travel health needs, and evaluating their adherence to recommended vaccines and oral therapies, satisfaction with the care provided, and their health status and management of health issues arising while travelling. Chart reviews will elicit descriptive quantitative data related to patients' travel medicine needs and adherence to recommended vaccinations and oral pharmacotherapy, followed by surveys containing open-ended qualitative questions to elicit overall patient satisfaction and the management of any health issues encountered during travel. Due to the nature of the study involving patients presenting to the clinic for a consultation, neither a control group nor blinding is possible.

A convenience sample of 100 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Receiving a pre-travel consultation at the Travel Health Network clinic in St. Albert, Alberta, Canada

Exclusion Criteria:

* Travellers with an expected return date after September 1, 2016
* Those receiving consultations as part of a group with the same itinerary (e.g., families, group vacations) will be asked to identify one member to participate in order to minimize repetition among participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals presenting for travel consultations at the Travel Health Network. No restrictions will be placed related to patient demographics, destinations, or travel itineraries; however, travellers with an expected return date after September 1, 2016 will be excluded, to ensure complete follow-up and data analysis within the proposed project time frame. A convenience sample of 100 patients will be consecutively enrolled .
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The proportion of recommended pre-travel vaccinations administered before departure according to chart review | Up to 7 months.
  From date of pre-travel consultation until the date of travel departure according to participant's planned itinerary, assessed up to September 2016.
The proportion of recommended pre-travel oral pharmacotherapies dispensed before departure by a community pharmacy according to electronic health record | Up to 7 months.
  From date of pre-travel consultation until the date of travel departure according to participant's planned itinerary, assessed up to September 2016.

SECONDARY OUTCOMES:
Average satisfaction (along 1-5 scale) with care provided elicited through an online survey post-travel | 1 week following return from travel according to participant's planned itinerary
Frequency of reason(s) for declining any recommended vaccines or medications according to participant self-report through an online survey | 1 week following return from travel according to participant's planned itinerary
  Response options: didn't feel I was at risk, cost, concern about vaccine ingredients or safety, other (specify)
Number of reports of any health issues over the course of travel according to participant self-report through an online survey | 1 week following return from travel according to participant's planned itinerary
  Response options: Traveller's diarrhea, Altitude sickness, Malaria, Fever (Dengue, Chikungunya), Respiratory illness, Other (specify)
Frequency of management strategies of any health issues over the course of travel according to participant self-report through an online survey | 1 week following return from travel according to participant's planned itinerary
  Response options: Nothing - it went away on its own, Took a non-prescription medication I had purchased before departure, Took a non-prescription medication I purchased while travelling, Called or emailed the Travel Health Network for advice, Searched the internet for guidance on how to manage it, Saw a physician while travelling, Saw a physician upon returning home, Other (specify)

CONTACTS AND LOCATIONS:
Locations (1):
- Travel Health Network, St. Albert, Alberta, Canada